CLINICAL TRIAL: NCT01546298
Title: Analysis of Immune Reactions Occurring Upon Administration of Patch Tests and Contact Dermatitis Affected Skin
Brief Title: Immune Reactions in Contact Dermatitis Affected Skin
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Collaborators: Washington University School of Medicine (Other); Tel Aviv University (Other)
Responsible Party: Sponsor
Other Study IDs: EGU-0757
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Allergic Contact Dermatitis
Keywords: Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Allergic Contact; Dermatitis, Contact | interventions — Patch Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patch tests of skin
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Patch tests — Patch tests for allergic reaction

SUMMARY:
This study hopes to improve the investigators understanding of how the immune system acts in allergic contact dermatitis. In order to reach this goal, normal volunteers, who are suspected of having allergic contact dermatitis, will be patch tested for the fifteen most common allergens. Then, biopsies will be taken of the skin at the sites where the there is a positive reaction to the allergen. Also, small biopsies will be taken from an area that received a patch but no allergen and an area that did not receive a patch to serve as controls. In a second stage of the study, volunteers will receive patches with the allergen to which they demonstrated an allergic response. More biopsies will be taken, over three designated time points. The biopsied skin samples will then be studied in a laboratory.

DETAILED DESCRIPTION:
Allergic contact dermatitis is a term for a skin reaction resulting from exposure to specific substances that come into contact with skin that is hypersensitive (allergic) to the substance. These substances are called "allergens." Some common allergens are nickel, rubber, dyes, poison ivy, poison oak and other related plants. These allergens do not cause a skin reaction in most individuals, but for some, once the skin becomes sensitive or allergic to the substance, any exposure to that specific allergen will produce a rash that may consist of redness, swelling and blisters. This rash may become worse with each exposure to the allergen. The skin reaction results from two phases. In the induction phase, initial exposure to the allergen occurs. The body recognizes the allergen as foreign and the immune system, which is the body's primary line of defense against infections and other things perceived as foreign to the body, mounts an immune response against the body, itself. During this immune response, cells specific to the allergen are activated. In the second phase, the elicitation phase, the skin is again exposed to the allergen and an immune response occurs, as the cells that are specific to the allergen attack the skin, leading to the rash. In order to diagnose allergic contact dermatitis, a clinician will discuss the materials that touch the patient's skin at work and home and perform patch tests. In a patch test, a very small amount of the suspected allergens are applied to the skin for a fixed time. After that designated time, the clinician will determine whether a reaction has occurred to the applied allergens. Currently, the main treatment for allergic contact dermatitis is avoidance of the allergen.

This study hopes to improve our understanding of how the immune system acts in allergic contact dermatitis. In order to reach this goal, normal volunteers, who are suspected of having allergic contact dermatitis, will be patch tested for the fifteen most common allergens. Then, biopsies will be taken of the skin at the sites where the there is a positive reaction to the allergen. Also, small biopsies will be taken from an area that received a patch but no allergen and an area that did not receive a patch to serve as controls. In a second stage of the study, volunteers will receive patches with the allergen to which they demonstrated an allergic response. More biopsies will be taken, over three designated time points. The biopsied skin samples will then be studied in a laboratory by methods such as immunohistochemistry and microarray analysis, which will help define the progression of the immune reaction in allergic contact dermatitis. The rationale for the study is to better understand how the immune system is activated to produce the rash of allergic contact dermatitis, so that treatments can target the cells that are involved in the activation.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-nursing female between 18 and 85 years of age
* Able to give verbal and written informed consent
* Must have a negative urine pregnancy test (for WOCBP).
* Must be suspected by clinician of having ACD (history or self-report of signs of ACD as defined as eczematous rash development with fragrances, use of non-gold or silver jewelry, use of hair dye, cosmetics) and/or a relevant food allergy (one of the allergens we will be testing)

Exclusion Criteria:

Subjects taking any of the following systemic or topical therapies within 2 weeks of enrollment: corticosteroids, immunosuppressants, and/or any other medications that may affect the outcome of the study

History of or suspected occupational allergies.

Subjects who are nursing mothers or pregnant

Hepatitis A, B, or C (self-reported)

Subjects who have active localized or systemic medical conditions that, in the opinion of the investigator, would preclude or make unsafe their participation in the study

Subjects who are unable to comply with study procedures, communicate effectively, cooperate with the investigator, or are unable to understand the study

Subjects who have been treated with an investigational device or drug within 30 days of enrollment

HIV positive as determined by self-reported history and/or a HIV POCT at screening

History, physical, social or lab findings suggestive of any medical or psychological condition that would, in the opinion of the PI, make the candidate ineligible for the study

Known anaphylactic reaction to food being tested in this study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Allergic Contact Dermatitis
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2012-12-14 (Actual); Study Completion 2012-12-14 (Actual)

PRIMARY OUTCOMES:
The response elicited by the allergen on relevant immune pathways as measured by cytokine levels in skin of IFNγ (Th1 pathway), IL-13 (Th2 pathway), IL-9 (Th9 pathway), IL-17 (Th17 pathway) and IL-22 (Th22 pathway). | 5 weeks
  The response elicited by the allergen on relevant immune pathways as measured by cytokine levels in skin of IFNγ (Th1 pathway), IL-13 (Th2 pathway), IL-9 (Th9 pathway), IL-17 (Th17 pathway) and IL-22 (Th22 pathway).

SECONDARY OUTCOMES:
Skin samples will be analyzed by immunohistochemistry for various cell types. | Day 2 and Day 7
  Skin samples will be analyzed by immunohistochemistry for various cell types including several T cell subsets (CD4+ vs CD8+ and Foxp3+ subsets), dendritic cells, natural killer cells, macrophages, B cells, and neutrophils. Expression of cytokine mRNAs in these samples will be used to assess Th1 (interferon-gamma), Th2 (IL-4, IL-13),Th17 (IL-17), and Th22 (IL-22) T cell activation.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Guttman, MD,PhD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided